CLINICAL TRIAL: NCT03183375
Title: An Open Label Randomized Controlled Trial to Evaluate the Efficacy and Safety of HYDROXYUREA in Management of Beta Thalassemia Patients in Karachi Pakistan
Brief Title: The Efficacy and Safety of HYDROXYUREA in Management of Beta Thalassemia Patients in Karachi Pakistan
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr.Saqib Hussain Ansari (Other)
Responsible Party: Sponsor-Investigator, Dr.Saqib Hussain Ansari, Principal Investigator, Omair Sana Foundation
Organization: Omair Sana Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERB0002
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Thalassemia, Beta
MeSH Terms: conditions — beta-Thalassemia | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: One is intervention arm which will be given investigational drug along with standard treatment and one will be control arm which will be given standard treatment only. Both groups will be assigned to only one treatment parallelly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxyurea arm (Experimental): This arm will be given investigational drug that is Hydroxyurea .This intervention will be given along with the standard treatment that is blood transfusion and iron chelation.
  Interventions: Drug: Hydroxyurea
- Standard arm (No Intervention): this arm will only receive the standard treatment which is blood transfusion and iron chelation

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea (starting from 10mg/kg/day with increasing dose by 2mg/kg/day until the desired response is achieved. The maximum dose given will be 20mg/kg/day)
  Arms: Hydroxyurea arm

SUMMARY:
Objectives

Primary objectives:

* To determine the efficacy of Hydroxyurea in the study participants.
* Hypothesis: The study will result in either maintenance or rise in hemoglobin as compared to the control treatment.

Secondary objectives:

* To determine the compliance of Hydroxyurea in study participants.
* To determine the safety of Hydroxyurea in the study participants. Design and Outcomes

An open label randomized controlled trial to test the efficacy and safety of Hydroxyurea on beta thalassemia major patients. It is a six months study. Findings of physical examination, vital sign variables, laboratory variables and ultrasound at baseline, during and end of the study will be listed. Schedule of intervention is mentioned in section 6.1. later in the protocol.

Interventions and Duration Hydroxyurea will be given to the participants in intervention arm along with the standard treatment if thalassemia (blood transfusion and iron chelation therapy) and the control arm will receive the standard treatment (blood transfusion and iron chelation therapy) only. Each participant will be followed up for 6 months after initiating the intervention. Intervention will be given for 6 months or until the participant withdraws from the study or due to any reason, the investigator stops the intervention.

Sample Size and Population This pilot study will be done on 100 patients initially. Stratified randomization will be done on the basis of presence of Xmn polymorphism. And the study population will be assigned to intervention or control arm randomly through a computer software (randomizer.org).

DETAILED DESCRIPTION:
Study Enrollment Procedures

* The study participants will be examined on the screening visit to assess their eligibility to participate. Each participant will consent in writing (Appendix I) to the screening process before the start of the examination and laboratory or radiology investigations. Screening log will be maintained to record this information.
* Parental consent (for minors age group < 18 years) will be obtained from a legal guardian accompanying the participant.
* The research unit will produce a computer generated sets of random allocations stratified on the basis of presence or absence of Xmn in advance of the start of the study. They will be then sealed in consecutively numbered opaque envelopes. The study participants will be randomly assigned to the investigation arm or control arm accordingly.

Storage and Accountability

All study drugs must be kept in a secure place under adequate storage conditions - protected from moisture and light and under required temperature (in refrigerator if required). Records of dispensing and returns will be maintained by the trial site (Omair Sana Foundation) in form of counts of tablets dispensed or returned. The subject must return all unused study medication for each treatment period to the trial center.

Statistical Analysis plan Intention to treat analysis Each participant will be analyzed in the group he was assigned to (investigational arm and control arm) at the time of study initiation rather than what he /she will take (drug orstandard treatment). Data will be entered and analyzed through statistical software SPSS version 17. Descriptive and inferential statistics will be analyzed. Descriptive statistics will be presented as means, standard deviations and ninety five percent confidence levels of the means for continuous variables and frequency and percentages for categorical variable.

Analysis per protocol patient:

Additional sensitivity analysis will be done as per protocol patient. Those participants will be analyzed who will receive at least 80% of the assigned intervention.

Inferential analysis: The mean difference in the efficacy and safety parameters from baseline to end will be reported along with p-value and ninety five percent confidence intervals. To find the difference, dependent T-test will be performed in case of normally distributed variables, Wilcoxan Signed Rank test for variables assuming non-parametric distribution and chi-square test of independence will be performed in case of categorical variables. The results will be displayed in form of graphs and tables. The results will be considered as statistically significant if p-value is less than 0.05 (level of significance).

Baseline characteristics: The demographic, background and baseline data and baseline characteristics of study participants will be presented descriptively. Protocol violations will be listed per participant, describing the nature of the violation. Participants failing to complete the study (as well as the times and reasons for discontinuation) will be displayed.

Analysis of Safety: Adverse Events, as reported throughout the course of the trial will be listed. Pre-, study and post-study findings of physical examination, vital sign variables, laboratory variables will be listed individually and summarized; values outside the normal range will be highlighted.

DATA COLLECTION AND QUALITY ASSURANCE Data Collection Forms Standard CRF (Appendix II) is designed for the data collection purpose. Data Management Database will be formed in order to record data from the folders for the trial patients.

Quality Assurance Data from the study will be collected in CRFs. Data editing will be performed at the trial center, comparing source and CRF entries.

During the study an independent monitor will visit the investigational site randomly without prior notification to confirm that the facilities remain acceptable, that the investigational team is adhering to the protocol and that data are being accurately recorded in the CRFs. Source data verification (a comparison of the data in the CRF with the participants' laboratory test results and other source documents) will also be performed.

Authorized representatives of the regulatory authority (e.g. IRB) may visit the center to perform inspections, including source data verification.

Clean File for the final database will be declared when all data have been entered and a quality check on a sample of the data has been performed. The database will be locked after Clean File has been declared and data extracted for statistical analysis.

Study committee meetings will be held as needed prior to or during the study. The medical, nursing and other research staff involved in the study will receive proper training on how to conduct the study and record the information according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with homozygous beta thalassemia major diagnosed on the basis of genetic mutation
* Beta thalassemia intermedia (patients carrying homozygous, heterozygous or compound heterozygous beta thalassemia genes) (HbS, HbE)
* Those patients who do not have baseline HbE suggestive of beta thalassemia, genetic mutations will be performed to confirm the diagnosis.
* Age: 6 months and onwards
* Gender: Either
* Able to understand study procedures and to comply with them for the entire length of the study.
* Provide written informed consent if aged 18 years and above and if minor that is below 18 years (Parental consent will be taken)

Exclusion Criteria:

* Chronic liver disease, renal failure, history of stroke
* Participants who have developed immune hemolytic anemia
* Spleenomegaly (liver and spleen >5 cm below coastal margin
* If allergic or sensitive to Hydroxyurea or its ingredients
* Patients on immunosuppressants including Azathiopine or any other drug causing bone marrow suppression, Hepatitis C treatment that may cause red cell suppression and NSAIDS
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
No. of participants who become responders or partial responders | 6 months
  The responders will be those who become transfusion independent (in those who were transfusion dependent before Hydroxyurea) or those who maintain or show 1-2 g/dl increase in Hb from baseline and partial responders will be those whose transfusion requirement decreases by atleast 50% as compared to baseline.

SECONDARY OUTCOMES:
The compliance of Hydroxyurea in study participants. | 6 months
  Compliance will be defined as actual number of tablets used/taken divided by the estimated number of tablets to be used/taken.
Number of participants with abnormal/deranged laboratory values | 6 months
  Participants with at least 1 of the following deranged laboratory values:
  * Deranged renal function (creatinine >2, Urea above normal range),
  * Liver function (SGPT 100 times more from baseline)
  * Neutropenia (neutrophil <1000)
  * Platelets < 50, 000
  * Deranged renal function (creatinine >2, Urea above normal range),
  * Liver function (SGPT 100 times more from baseline)
  * Neutropenia (neutrophil <1000)
  * Platelets < 50, 000 Deranged renal function (creatinine >2, Urea above normal range), Liver function (SGPT 100 times more from baseline),Neutropenia (neutrophil <1000),Platelets < 50, 000
No. of participants with severe adverse events related to the intervention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Saqib H Ansari, MBBS, DCH, DPGN, Mphil, PhD, Principal Investigator — Omair Sana Foundation
Locations (1):
- Omair Sana Foundation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No